CLINICAL TRIAL: NCT02265614
Title: Preimplantation Genetic Screening (PGS) Using Microarray Technique: Method to Select the Embryo With the Greatest Chance for Successful Implantation During in Vitro Fertilization in Couples With a History of Unsuccessful IVF Attempts
Brief Title: PGS Using Microarray in IVF Patients With Repeated Implantation Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IVF Research Sweden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IVFResearch
Record Dates: First submitted 2014-10-10; First posted 2014-10-16 (Estimated); Last update posted 2014-10-20 (Estimated); Status verified 2014-10

CONDITIONS: Infertility
Keywords: PGS; blastocyst; human; IVF; vitrification; single embryo transfer
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PGS (Experimental): blastocyst biopsy and chromosomal analysis
  Interventions: Genetic: PGS
- control (No Intervention): regular IVF

INTERVENTIONS:
Genetic: PGS
  Arms: PGS

SUMMARY:
This project intends to use preimplantation genetic screening (PGS) with the microarray technique to determine the chromosome composition of fertilized eggs, so that only chromosomally normal embryos are transferred during IVF. The purpose is to increase the probability of pregnancy and childbirth among couples with a history of repeated unsuccessful IVF attempts.

DETAILED DESCRIPTION:
Background In vitro fertilization (IVF) is the most important method to remedy infertility, whether the cause is the male or the female, or when the cause is unknown. Treatment usually involves the transfer to the uterus of a fertilized egg (embryo) that has been cultured for 2-5 days. To select the embryo with the best chance of successful implantation into the endometrium, microscopic evaluation is currently used to grade embryonic cell division, cellular appearance, and other factors. But this method is incomplete because it cannot determine the functional properties of the embryo, or whether it is genetically normal. It is known that couples with a history of multiple unsuccessful IVF treatments produce a large number of embryos that have an abnormal number of chromosomes (aneuploidy), which is also common in women over age 38.

This project intends to use preimplantation genetic screening (PGS) with the microarray technique to determine the chromosome composition of fertilized eggs, so that only chromosomally normal embryos are transferred during IVF. The purpose is to increase the probability of pregnancy and childbirth among couples with a history of repeated unsuccessful IVF attempts. We have previously conducted a prospective randomized study with a similar question (Ö 612-02) on a target group of older women (>38 years) using sampling (biopsy) of the embryo on day 3 of culture, followed by analysis of seven chromosome pairs using the FISH technique. The results of the study showed no improvement in pregnancy outcome . The reasons are probably 1) to begin with, normal eggs are infrequent in this target group; 2) the biopsy was performed on day 3 when the embryo is at a sensitive stage; and 3) only 7 out of a total of 23 chromosome pairs could be analyzed.

Methodological developments in the field have been rapid, and current technology allows for better identification of normal embryos compared with the previous study.

* We know that the embryo is less sensitive when a biopsy is carried out on day 5 (of the blastocyst stage) instead of day 3.
* In blastocyst biopsy, more cells are removed for diagnosis than on a day 3 biopsy (thereby increasing the reliability of the analysis).
* Blastocyst biopsy involves removal of fewer cells on a percentage basis (3-5%) from the total cell mass of the blastocyst compared with the previously used day 3 biopsy, which involved removal of up to 25% of the total number of cells.
* Blastocysts have a higher implantation rate than day 3 embryos.
* Array Comparative Genomic Hybridization (aCGH) can now be used with great precision to analyze all chromosomes using commercial quality-controlled kits.
* Cryopreservation with vitrification of blastocysts is currently a highly successful technique that allows the analysis to be conducted without being pressed for time.

In addition, we will turn to a patient group consisting of women with a proven normal-good ovarian reserve. In the previous study involving women >38 years, the ovarian reserve was generally poor.

The preparatory work for the Genetic Integrity Act stated that PGS should "be reserved for clearly defined research projects approved in an ethical review by an ethics committee." This restriction was imposed because the state of knowledge about PGS at that time was very limited. More experience from research projects on PGS was considered necessary to determine whether PGS could be used in clinical practice. The above mentioned preparatory work for the Genetic Integrity Act also states that PGS "may become an important tool to increase chances of pregnancy in conjunction with IVF treatment ...". In this project, we intend to investigate whether it is possible to increase the chance of pregnancy and childbirth among couples who have undergone several previous failed IVF attempts. Our hypothesis is based on the assumption that an incorrect number of chromosomes is often the underlying cause of failed implantation or miscarriage. To increase the chances of establishing a pregnancy that leads to childbirth, we are conducting a chromosome analysis on the embryos of couples to ensure that only embryos with a normal chromosome set are transferred to the woman.

Question Can the probability of pregnancy and childbirth in couples with several previous failed IVF attempts increase if a normal chromosome set can be ensured in the embryo before it is transferred? As a control, we will compare the results of IVF attempts where only light microscopic evaluation is performed.

Primary endpoint: Delivery per randomized patient Secondary endpoints: Cumulative pregnancy rate including later transfer of remaining vitrified blastocysts (higher rate expected in study group). Miscarriage rate during the first 18 weeks of pregnancy (lower rate expected in study group).

Methods and materials Patients Couples with a history of at least three unsuccessful IVF attempts, in which the woman is a maximum of 39 years of age, will be invited in conjunction with their consultation for a new IVF treatment at any of IVF Sweden clinics to participate in the study, provided that they meet the inclusion criteria (including expected normal response to hormone stimulation with 8-10 eggs). The women who agree to participate in the study will be randomized (by computer) to either the biopsy or the control group the day after collection of oocytes if they have at least 5 fertilized eggs (current procedure for culture on day 5).

Inclusion criteria: Couples who meet the criteria for IVF treatment and who have a history of at least three previous IVF cycles including embryo transfer without delivery. The woman may be a maximum of 39 years old when the study is carried out and must have a normal-good ovarian reserve ( at least 12 antral follicles). Her partner must be able to provide a semen sample containing live sperm. Women included in the study will not participate in any other research project.

Exclusion criteria: Myoma, or other uterine lesions judged to affect implantation. Nonspecific cysts that are not considered to be functional. Endometrium >3 cm.

Randomization

Randomization will take place on day 1 if the couple meets the requirements established for culture to the blastocyst stage (at least 5 normally fertilized oocytes). The on-line randomization program (computerized) will balance the following parameters:

* Age
* Number of oocytes retrieved

Furthermore at the time of randomization, the randomization program will take into account that a multicenter study is involved to avoid bias.

IVF treatment Hormone stimulation, ultrasound checks, collection of oocytes, and fertilization will follow standard procedure. For women in the control group, all expanded blastocysts will be cryopreserved (vitrified) day 5-6 for later transfer. For women randomized to PGS, cells (trophectoderm cells in the outer cell layer of the embryo) will be biopsied on day 5-6 after which all biopsied blastocysts will be vitrified. If the analysis shows a normal chromosome set, the blastocyst will be thawed and transferred during the next menstrual cycle.

Biopsy and cell lysis The biopsy is carried out by making a hole in the shell of the blastocyst (zona pellucida) using laser technology and special biopsy equipment and removing 2-5 cells from the outer cell mass (trophoblast cells). The cells are transferred to a test tube containing PBS solution. An extraction solution is added to lyse the cells, and the DNA is released into the solution.

Optimization of genome amplification To optimize the protocol for cell lysis and whole genome amplification, cells from an embryonic stem cell line with trisomy 13 as well as from a normal karyotype will be used. Three, four and five cells respectively will be pipetted into PCR tubes. The entire aCGH protocol (see below) will be run on these cells (at least 50 tubes), and the results will be evaluated. This approach will provide us with an idea of the sensitivity of the method and how often we fail to obtain results due to unsuccessful amplification. Contamination in the system, if any, will also be revealed.

Array Comparative Genomic Hybridization (aCGH) Reagent for amplification (copying) of the DNA is added to the DNA extract. Amplification is carried out in several steps using a technique called "Polymerase Chain Reaction" (PCR). This process requires great accuracy and special laboratory facilities so that foreign DNA does not contaminate the sample. Contamination at this step could lead to a misdiagnosis of the chromosome constitution of the embryos. The amplified DNA is then labeled with a fluorescent molecule which causes the DNA to fluoresce green under UV illumination. Similarly, normal control DNA is labeled with a molecule that fluoresces red under UV illumination. Amplified fluorescently labeled DNA is mixed with an equal volume of normal fluorescently labeled control DNA. This DNA mixture is applied to test surfaces with specific DNA sequences. These DNA sequences are carefully selected and placed on the test surfaces in long arrays in a specific order, which means that DNA from all chromosome arms are represented on the test surface at specific locations. During the hybridization step, the DNA in the DNA mixture will compete for binding to the DNA on the test surface. If there are equal amounts of amplified DNA (green) and control DNA (red), then an equal amount of DNA from both fractions will bind to the test surface. After hybridization, when the test surface is illuminated with UV light, the green and red fluorescence will be equally intense, resulting in an orange color (mixture with equal portions of red and green color). However, if there is an excess of DNA from a given chromosome in the embryo (e.g., trisomy), more DNA sequences from this chromosome will bind to the test surface, resulting in an excess of green fluorescence in the area on the test surface containing the DNA sequences from the relevant chromosome. Similarly, loss of a chromosome in an embryo results in a shortage of the corresponding DNA in the amplified fraction, causing more control DNA sequences (red) to bind to the test surface. Test areas are scanned and results processed automatically in a computerized scanner.

Grading of embryos:

Evaluation and grading of the blastocysts will be done in accordance with accepted classification according to Gardner in which degree of expansion, cell density, and number of cells in the inner cell mass (IC) and in the trophectoderm (TE) are assessed. All blastocysts in the control group will be vitrified for later transfer. A similar evaluation will be carried out in the biopsy group prior to biopsy. Following biopsy, all biopsied blastocysts will be vitrified.

In the group in which the biopsy is conducted, microarray analysis will be carried out. Transfer is done during the natural menstrual cycle 5 days after ovulation. Women with hormonal disruption require mild hormonal stimulation prior to transfer of the vitrified/warmed blastocyst.

Vitrification After the blastocysts have been biopsied, they will be vitrified and subsequently thawed according to well established protocol at the clinics.

Follow-up The primary endpoint is birth per randomized patient. Secondary endpoints are cumulative pregnancy rate, since extra cryopreserved blastocysts (if any) are also transferred, and miscarriage rate during the first 18 weeks of pregnancy (lower rate expected in study group). We plan to create a Data Safety Monitoring Board (DSMB) consisting of independent external experts when half the study has been completed.

Follow up of all pregnancies and childbirths will be carried out according to current procedure within IVF.

Statistics Power analysis has shown that to detect a significant difference in pregnancy outcomes from the estimated 15% in the control group to 40% in the PGS group requires 112 patients (alpha=0.8; Beta=0.20). An estimated attrition rate of about 10% and the planned DSMB analysis mean that 130 patients should be recruited. The DSMB will monitor the study and provide periodic advice on whether we should continue the study. The DSMB analysis will give 3 recommendations: (1) continue the study as planned, (2) stop the study if the difference between the groups is less than 15 %, (3) continue the study with a larger sample size. When the difference between the groups are 20 % or greater the study can be continued with a larger sample size (73 patients in each group The DSMB analysis will advice to continue or stop the study (due to highly significant effect, negative effect or low conditional power. DSMB can evaluate both live birth and ongoing pregnancy and weigh all information when they give the recommendation. The DSMB will consist of specialists who are experienced in this field. Statistical calculations will be carried out according to intention-to-treat (ITT), as well as per protocol . ITT are all randomized patients, having at least 5 fertilized oocytes on day 1. Some patients are likely to have no transfer due to the lack of blastocysts,or technical problems relating to vitrification/warming etc. Therefore, analysis will also be done per protocol. Logistic regression will be used in the statistical calculations and include the stratification variables.

ELIGIBILITY:
Inclusion Criteria:

* Couples who meet the criteria for IVF treatment and who have a history of at least three previous IVF cycles including embryo transfer without delivery.
* The woman may be a maximum of 39 years old when the study is carried out and must have a normal-good ovarian reserve (at least 12 antral follicles).
* Her partner must be able to provide a semen sample containing live sperm.
* Women included in the study will not participate in any other research project.

Exclusion Criteria:

* Myoma, or other uterine lesions judged to affect implantation.
* Nonspecific cysts that are not considered to be functional.
* Endometrium >3 cm.

Ages: 25 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 130 (Estimated)
Dates: Start 2014-08; Primary Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
ongoing pregnancy per randomized patient | 2 years

SECONDARY OUTCOMES:
cumulative pregnancy rate, | 3 years
miscarriage rate during the first 18 weeks of pregnancy | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Fertilitetscentrum AB, Gothenburg, Sweden